CLINICAL TRIAL: NCT00370357
Title: A Phase 1, Placebo Controlled Study of the Safety of 3% w/w SPL7013 Gel, Administered to the Penis of Healthy Male Volunteers Once Daily for Seven Days
Brief Title: SPL7013 Gel - Male Tolerance Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Starpharma Pty Ltd (Industry)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Marcus Chen MD, Melbourne Sexual Health Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: SPL7013-002
Record Dates: First submitted 2006-08-30; First posted 2006-08-31 (Estimated); Last update posted 2008-01-16 (Estimated); Status verified 2008-01

CONDITIONS: Human Immunodeficiency Virus (HIV)
Keywords: Microbicide; SPL7013; VivaGel
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — astodrimer

INTERVENTIONS:
Drug: 3% w/w SPL7013 Gel (VivaGel™)

SUMMARY:
The purpose of this study is to determine if SPL7013 Gel (VivaGel™) is safe when applied topically once a day for seven consecutive days to the shaft and glans of the penis in healthy male volunteers. The study will compare the safety of SPL7013 Gel on the penile epithelium and urethral mucosa to the safety of a placebo gel. The study will also assess the systemic safety of SPL7013 Gel, systemic absorption of the active ingredient of SPL7013 Gel, and the acceptability of the study products to the male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent
* Healthy males aged 18 years or older
* HIV negative
* Reports vaginal intercourse in the past 12 months
* Agrees to abstain from vaginal, anal (receptive and insertive) and oral sexual intercourse, and agrees to refrain from masturbation during the 7 days of product use until after the End-of-Treatment (Day 7) study visit

Exclusion Criteria:

* Known or suspected allergy to any component of the study products or similar ingredients in other products
* History of significant drug reaction or allergy
* Recent history (within 12 months) or presence at screening of contact dermatitis or other dermatological condition
* Recent history (within three months of Screening) of a sexually transmitted infection (STI)
* Current signs or symptoms of UTI and/or STI at Screening or Baseline
* Positive urine leukocyte esterase test (≥ trace)
* Biochemical and/or haematological parameters outside the laboratory's normal reference ranges at Screening
* Evidence of genital piercing, ulceration, genital dermatoses, tinea cruris or other dermatological condition of the genitalia or upper thighs
* Genital pain or discomfort at Screening or Baseline
* Any other abnormal finding on physical examination or other medical condition

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36
Dates: Start 2006-08; Primary Completion 2007-02 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Participant reports of genital pain, genital burning, penile itching, penile rash, penile ulceration or other genital symptoms
Erythema, vesiculation, bullous reaction, ulceration or other genital findings of the penile shaft, foreskin, glans or meatus as observed by visual examination

SECONDARY OUTCOMES:
All other adverse events
Laboratory abnormalities
Plasma concentrations of SPL7013
Expectations and experiences of the study products described by participant interviews

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Chen, MD, PhD, Principal Investigator — Melbourne Sexual Health Centre
Locations (1):
- Melbourne Sexual Health Centre, Carlton, Victoria, Australia